CLINICAL TRIAL: NCT05138744
Title: Behavioral Activation for Depression Through Virtual Reality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMA1
Record Dates: First submitted 2021-07-26; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Single case design (multiple baselines)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality treatment (Experimental): Use of google maps with virtual reality to virtually situate the participants into scenarios that are motivating for them (i.e., the beach, a mountain, a park, etc.) at their choice.
  Interventions: Other: Behavioral activation using virtual reality

INTERVENTIONS:
Other: Behavioral activation using virtual reality — The investigators will encourage behavioral activation (increase in the number and time of conducted activities) situating the person in motivating situations using virtual reality

SUMMARY:
Evaluate the effectiveness of a brief, virtual reality intervention for depressed mood

ELIGIBILITY:
Inclusion Criteria:

* Patient Health Questionnaire - 9 (measure of depression) over 9
* Positive and Negative Affect Schedule (measure of positive and negative affect): positive affect score below 24
* Age over 18 years
* Signs informed consent

Exclusion Criteria:

* Completes more than 20% of evaluations retrospectively (not the day they are assigned)
* Has a severe mental health disorder as evaluated with the MINI International Neuropsychiatric Interview
* Does not sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-12-05 (Estimated); Primary Completion 2022-01-22 (Estimated); Study Completion 2022-02-20 (Estimated)

PRIMARY OUTCOMES:
Change in Behavioral activation | Change through study completion, an average of 31 days. The outcome will be evaluated daily (at 9pm) during 31 days. Changes will be investigated from baseline to posttreatment using all corresponding time points (baseline vs posttreatment)
  In a scale from 0 (not at all) to 6 (completely), "to what extent were you satisfied with what you did today?"

SECONDARY OUTCOMES:
Change in Mood | Change through study completion, an average of 31 days. The outcome will be evaluated daily (at 9pm) during 31 days. Changes will be investigated from baseline to posttreatment using all corresponding time points (baseline to posttreatment)
  In a scale from 0 (completely sad) to 100 (completely happy), "how did you feel today?"
Change in Depression | Change through study completion, an average of 31 days.. The outcome will be evaluated daily (at 9pm) during 31 days. Changes will be investigated from baseline to posttreatment using all corresponding time points (baseline to posttreatment)
  In a scale from 0 (not at all) to 3 (completely), "how was your level of depression today?"
Change in Positive affect | Change through study completion, an average of 31 days.. The outcome will be evaluated daily (at 9pm) during 31 days. Changes will be investigated from baseline to posttreatment using all corresponding time points (baseline to posttreatment)
  In a scale from 1 (not at all) to 5 (completely), "how was your positive affect today?"
Change in Negative affect | Change through study completion, an average of 31 days.. The outcome will be evaluated daily (at 9pm) during 31 days. Changes will be investigated from baseline to posttreatment using all corresponding time points (baseline to posttreatment)
  In a scale from 1 (not at all) to 5 (completely), "how was your negative affect today?"
Change in Activity level | Change through study completion, an average of 31 days.. The outcome will be evaluated daily (at 9pm) during 31 days. Changes will be investigated from baseline to posttreatment using all corresponding time points (baseline to posttreatment)
  In a scale from 0 (minimum) to 100 (maximum), "what was your activity level today?"

IPD SHARING:
Plan to Share IPD: No
Data will be anonymized and will only be shared upon reasonable request without identifying information